CLINICAL TRIAL: NCT00163241
Title: A Double-Blind, Placebo-Controlled, Randomized 24-Month Study, Assessing The Effect Of Celecoxib (Celebrex) Long Term Treatment On Hip Osteoarthritis (OA) Progression OSCARE
Brief Title: Effect Of Celecoxib On Hip Osteoarthritis (OA) Progression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see detailed description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A3191068
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
Objectives of the study:

Primary: Assess the ability of a continuous treatment of celecoxib 200 mg versus placebo administered once daily (QD) for 24 months in slowing disease progression as assessed radiographically in subjects with osteoarthritis (OA) of the hipSecondary:Assess the ability of a continuous treatment of celecoxib 200 mg versus placebo administered QD for 24 months in treating disease signs and symptoms in subjects with OA of the hip.Evaluate the ability of a continuous 24-month intake of celecoxib 200 mg QD versus placebo to reduce number of subjects eligible for hip replacement according to the investigator.Evaluate the tolerability and safety of a continuous 24-month intake of celecoxib 200 mg QD versus placebo in subjects with OA of the hip.

DETAILED DESCRIPTION:
The study was terminated on 19 January 2006, prematurely, as a result of low enrollment Safety concerns did not lead to the decision to terminate this study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 50 years of age or older.
* If the subject is a female and of childbearing potential, or less than 2 years post-menopausal, she must have been using adequate contraception during her last menses and will use adequate contraception during the study, is not lactating, and has had a negative urine pregnancy test within 24 hours prior to receiving the first dose of study medication. Women less than two years post-menopausal are considered of childbearing potential for the purposes of this study.
* The subject is diagnosed as having OA of the hip as defined by the American College of Rheumatology (ACR) criteria (see Appendix B)
* The subject has symptomatic OA, as defined by the presence of daily hip pain for at least 1 month (not necessarily continuously) during the 2 months prior to screening visit.
* The subject has hip pain of > or equal to 3 and < or equal to 9 on a 10-point Visual Numerical Scale (VNS) in the index hip.
* Subjects with OA of the knee associated with OA of the hip will be included provided knee OA pain intensity is inferior to hip's one and no knee surgery is expected during the study.
* Subjects are functional class I, II or III according to the Steinbrocker criteria (see Appendix C).
* The subject is eligible for pharmacologic treatment to control arthritis symptoms.
* The subject has provided written informed consent before undergoing any study procedures.

Exclusion Criteria:

* Bilateral hip OA with contralateral hip more severe symptomatically or radiologically than the index hip.
* The subject has evidence of secondary hip OA.
* Septic arthritis
* Systemic or local inflammatory joint disease (e.g. psoriatic arthritis, spondylarthropathy, systemic lupus erythematosus, etc.)
* Gout
* Recurrent episode of pseudogout
* Paget's disease
* Articular fracture
* Ochronosis
* Acromegaly
* Haemochromatosis
* Wilson's disease
* Primary osteochondromatosis
* Osteonecrosis
* Slipped Capital Femoral Epiphysis (SCFE)
* The subject has a concomitant inflammatory rheumatic condition, which may interfere with the assessment of OA, or acute joint trauma at the index hip.
* The subject has received oral, intramuscular, intravenous, or soft tissue injection of corticosteroids within 4 weeks prior to the screening visit.
* The subject has received an intra-articular injection of corticosteroids or hyaluronic acid in the index hip within 12 weeks prior to the screening visit.
* The subject has received diacerein, chondroitin sulfate, glucosamine sulfate, doxycycline or avocado/soybean unsaponifiables within 12 weeks prior to the screening visit.
* Arthroscopy or a corrective surgery of the index hip has been performed.
* Arthroscopy or a corrective surgery of the contralateral hip has been performed within the 6 months prior to the screening visit .
* Total replacement of the contralateral hip joint was performed within 6 months prior to the screening visit.
* The subject is felt to require hip arthroplasty by the investigator at screening visit.
* The subject has an active malignancy of any type. Subjects who have a history of basal cell carcinoma that has been successfully treated are acceptable. Subjects with a history of other malignancies that have been successfully treated and who have no evidence of recurrence for at least 5 years before study are also acceptable.
* The subject has been diagnosed as having or has been treated for esophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to the screening visit.
* The subject has a history of recurrent ulceration or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a chronic or acute renal or hepatic disorder, a significant coagulation defect, or any other condition, which in the investigator's opinion might preclude use of NSAIDs.
* The subject has a history of intolerance to paracetamol, opioids and tramadol such that it is felt that an adequate non-anti-inflammatory rescue analgesic regimen cannot be safely prescribed, or has a history of alcohol or substance abuse.
* The subject has known hypersensitivity to celecoxib, demonstrated allergic-type reactions to sulfonamides, experienced asthma, urticaria or allergic-type reactions after taking sulfonamides, aspirin (acetylsalicylic acid [ASA]), lactose or NSAIDs.
* The subject has been diagnosed as having or has been treated for gastrointestinal bleeding within 30 days before the screening visit.
* The subject has previously been admitted to this study.
* The subject has a likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (see Section 9 "Concomitant therapy").
* The subject has severe disease, likely to jeopardize the planned completion of the study
* The subject has abnormal baseline findings and or any other condition, which, in the investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* The subject is not literate in French nor English or is unable according to the investigator to answer questions.
* The subject has received any investigational drug within 30 days prior to the screening visit.
* The subject has a history of myocardial infarction, unstable angina, ischemic or hemorrhagic stroke, transient ischemic attack, previous revascularization procedure to coronary, carotid, cerebral, renal, aortic or peripheral arterial vasculature.
* The subject has congestive heart failure (Class II-IV).
* The subject is using aspirin, including low dose aspirin.
* The subject is using other antiplatelet agents (ticlopidine, clopidogrel, dipyridamole).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666
Dates: Start 2004-06; Study Completion 2006-01

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in the minimal JSW of the index hip during the 24-month follow up, compared to baseline. This endpoint will be expressed as the proportion of subjects achieving a 0.5 mm decrease in JSW on a radiograph and

SECONDARY OUTCOMES:
Number of days with rescue medication usage by drug category: paracetamol /paracetamol combination products, opioid/opioid combination products, celecoxib and other (e.g., propoxyphene) WOMAC subscales: pain and function (in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (110):
- Canada (8):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
  - Pfizer Investigational Site, Trois-Revieres, Quebec
  - Pfizer Investigational Site, St. John's
- France (102):
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Antibes
  - Pfizer Investigational Site, Arles
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Bagnols-sur-Cèze
  - Pfizer Investigational Site, Beauvais
  - Pfizer Investigational Site, Belfort
  - Pfizer Investigational Site, Boulogne-sur-Mer
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Cahors
  - Pfizer Investigational Site, Cannes La Boca
  - Pfizer Investigational Site, Castelnaudary
  - Pfizer Investigational Site, Chateuauroux
  - Pfizer Investigational Site, Chaumont
  - Pfizer Investigational Site, Cherbourg
  - Pfizer Investigational Site, Clamart
  - Pfizer Investigational Site, Clichy
  - Pfizer Investigational Site, Colmar
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, Cornebarrieu
  - Pfizer Investigational Site, Courbevoie
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Dax
  - Pfizer Investigational Site, Digne-les-Bains
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Épernay
  - Pfizer Investigational Site, Firminy
  - Pfizer Investigational Site, Fontainebleau
  - Pfizer Investigational Site, Gardanne
  - Pfizer Investigational Site, Gonesse
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Issy-les-Moulineaux
  - Pfizer Investigational Site, Ivry-sur-Seine
  - Pfizer Investigational Site, Jonzac
  - Pfizer Investigational Site, Joué-lès-Tours
  - Pfizer Investigational Site, L'Aigle
  - Pfizer Investigational Site, L'Union
  - Pfizer Investigational Site, La Celle-Saint-Cloud
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, Landivisiau
  - Pfizer Investigational Site, Langon
  - Pfizer Investigational Site, Laval
  - Pfizer Investigational Site, Le Perreus Sur Marne
  - Pfizer Investigational Site, Le Petit-Quevilly
  - Pfizer Investigational Site, Les Angles
  - Pfizer Investigational Site, Libourne
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Lisieux
  - Pfizer Investigational Site, Lunel
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Maisons-Alfort
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Martigues
  - Pfizer Investigational Site, Montgeron
  - Pfizer Investigational Site, Montigny-le-Bretonneux
  - Pfizer Investigational Site, Montluçon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Moulins
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Naucelle
  - Pfizer Investigational Site, Neufchâteau
  - Pfizer Investigational Site, Nevers
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Nogent-le-Rotrou
  - Pfizer Investigational Site, Obernai
  - Pfizer Investigational Site, Orléans
  - Pfizer Investigational Site, Orly
  - Pfizer Investigational Site, Ormesson-sur-Marne
  - Pfizer Investigational Site, Orthez
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Puteaux
  - Pfizer Investigational Site, Quimper
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rodez
  - Pfizer Investigational Site, Saint Afrique
  - Pfizer Investigational Site, Saint Genevvieve Des Bois
  - Pfizer Investigational Site, Saint Giron
  - Pfizer Investigational Site, Saint Maxime
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Saint-Jacques-de-la-Lande
  - Pfizer Investigational Site, Saint-Lô
  - Pfizer Investigational Site, Saint-Pierre-de-Coutances
  - Pfizer Investigational Site, Saint-Quentin
  - Pfizer Investigational Site, Sartrouville
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Thionville
  - Pfizer Investigational Site, Thonon-les-Bains
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tourcoing
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Valence
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Vence
  - Pfizer Investigational Site, Versailles
  - Pfizer Investigational Site, Villeneuve-sur-Lot
  - Pfizer Investigational Site, Villeurbanne
  - Pfizer Investigational Site, Vitré
  - Pfizer Investigational Site, Vitrolles

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191068&StudyName=Effect+Of+Celecoxib+On+Hip+Osteoarthritis+%28OA%29+Progression